CLINICAL TRIAL: NCT03930628
Title: Limb-Girdle Muscular Dystrophy Type 2I in Norway - a Cohort Study
Brief Title: Limb-Girdle Muscular Dystrophy Type 2I in Norway
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); Norwegian Muscle Disease Association (FFM) (Unknown); Norwegian National Advisory Unit on Rare Disorders (NKSD) (Unknown); Norwegian Competence Center for Sleep Disorders (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018/1968(REK)
Record Dates: First submitted 2019-04-15; First posted 2019-04-29 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Limb Girdle Muscular Dystrophy, Type 2I; Limb Girdle Muscular Dystrophy; Muscular Dystrophies; Limb Girdle Muscular Dystrophy R9 FKRP-related
MeSH Terms: conditions — Muscular Dystrophy, Limb-Girdle, Type 2I; Muscular Dystrophies, Limb-Girdle; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Key goals are to establish the natural history of limb-girdle muscular dystrophy type 2I (LGMD 2I) and identify feasible and sensitive tools and biomarkers to measure disease affection and progression, determine the Norwegian LGMD 2I prevalence, carrier frequency and genotypes, and to assess health-related quality of life in the Norwegian LGMD 2I population.

Main aims are to facilitate future clinical trials and contribute to good clinical practice with suitable methodology and to complete health and social care in order to optimize the function and quality of daily living of the patient group.

DETAILED DESCRIPTION:
A single-center study with Norwegian nationwide enrollment. Data is based on questionnaires, patient journals, clinical examination, a set of functional tests and biomarkers, and patient reported outcomes. Clinical/ paraclinical tests are repeated after 2-years in order to measure disease progression. Both skeletal muscle, heart and respiratory function will be examined. At baseline there will also be performed a sleep study in order to find if they are prone to sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Genetical confirmed limb-girdle muscular dystrophy type 2I in Norway
* Live in Norway
* Written consent

Exclusion Criteria:

* Children < 16 years are excluded from the assessment of quality of life and from the clinical/paraclinical part, but may contribute with information through questionnaires and patient journal.

The study of prevalence and genotypes is anonymous and consent independent and will include everyone that is genetically LGMD 2I-confirmed in Norway.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of limb-girdle muscular dystrophy type 2I genetically confirmed in Norway and who live in Norway.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Echo intensity of muscles | Baseline and 2 years
  Change in echo intensity at a defined cross-sectional level in muscles in limbs, musculus rectus abdominis and paraspinal muscles from baseline at 2 years. Echo intensity is measured as grayscale pixels ranging from 0 (black) to 255 (white) through histogram analysis by an ultrasound software program. It calculates the mean value from the superficial 1/3 of a manually selected region of interest in three consecutive images from same location. Increase in echo intensity indicates increase in pathology.
Muscle thickness | Baseline and 2 years
  Using ultrasound to measure changes in muscle thickness at a defined cross-sectional level in muscles in limbs, musculus rectus abdominis and paraspinal muscles from baseline at 2 years.
Age at important disease stages | Retrospective data collection at baseline
  Document the variation in age of onset, age of loss of walking ability, age of established cardiac failure and age of established respiratory failure.
Rate of symptom progression | Retrospective data collection at baseline
  Document the variation in time from disease onset to loss of walking ability
Prevalence of recognized cardiomyopathy | Retrospective data collection at baseline
  The percentage of females and males with recognized cardiomyopathy
Prevalence of initiated ventilation support | Retrospective data collection at baseline
  The percentage of female and males that have initiated ventilation support.
Motor task performance | Baseline and 2 years
  Using the standardised scoring instrument "Motor Function Measure for neuromuscular diseases" (MFM) to measure the ability to perform 32 different motor tasks. The individual item score ranges from 0 (cannot initiate the task) to 3 (performs fully and normally). The items are divided into 3 domains: 1) Standing and transfers (13 tasks), 2) Axial and proximal motor function (12 tasks), 3) Distal motor function (7 tasks). The 3 domains give rise to 3 subscores. Both subscores and total score (0-96 points) will be measured. Baseline and changes from baseline at two years.
Disease-specific health-related quality of life (HRQOL) | Baseline, at 6 months, 1 year
  Using the "Individualized Neuromuscular Quality of Life" (INQOL)-questionnaire to measure the burden of disease. It consists of 45 items. Each item is graded by a 7-point Likert scale (0-6/1-7).The 45 items make up 3 dimensions/domains: muscular symptoms, effects on life-domains (activities, independence, emotions, body image, social relationships) and effects of treatment. The 3 domains are together subdivided into 11 subdimensions, each with its own subscale. In addition there is a QOL-score which is a composite score from the "Life-domain". The scores range from 0-100 and are determined by the item responses and a weighting algorithm. The higher the scores, the more negative impact. Both subscales and QOL-score will be determined - at baseline and changes from baseline at 6 months, 1 year and 2 years.
Echocardiography strain speckle-tracking | Baseline and 2 years
  Measure cardiac function at baseline and changes from baseline at 2 years
Nocturnal arterial carbon dioxide (CO2)-level | Baseline
  Monitor transcutaneous CO2 during sleep at baseline.
MRI | At 2 years
  Muscle MRI lower limbs

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | Baseline (2 tests with 1 day interval) and two years (2 tests with 1 day interval)
  Walk distance in 6 minutes, Borgs scale for dyspnoea and fatigue pre and post test, and for self-reported exertion. Changes from baseline in 6MWT at 2 years
4-step stair climb test | Baseline and 2 years
  Changes from baseline in time to ascend and to descend a 4-steps stair at two years
Level of motor independence: "Vignos Grade" | Baseline and 2 years
  Using "Vignos grade" to score level of motor independence. The score ranges from 1 (walk and climb without assistance) to 10 (confined to bed).
Upper limb movement ability: "Brooks Grade" | Baseline and 2 years
  Using "Brooks Grade" to score the ability to raise arms above the head, ranging from 1 (normal: full abduction until the hands touch above the head) to 6 (cannot raise hands to mouth and has no useful function of hands). Baseline and changes from baseline at two years.
Hand held dynamometry | Baseline and 2 years
  Changes from baseline in muscular strength in the limbs at two years
Manual Muscular Testing (MMT) | Baseline and 2 years
  Changes from baseline in muscular strength in the limbs at two years
General health-related quality of life | Baseline, 6 months, 1 year
  Using the Norwegian translation of general HRQOL-instrument "Short Form Health Survey" (SF-36). It is a questionnaire with 36 questions (items) investigating 8 domains/dimensions (physical function, physical role limitations, emotional role limitations, social functioning, bodily pain, general health perceptions, vitality, mental health). The 8 domain scores will be determined. The scores range from 0-100 and are based on item-responses and weighting algorithm. High score stands for good health. Measure at baseline and changes from baseline at 6 months, 1 year and 2 years.
Plethysmography | Baseline and 2 years
  Lung volumes at baseline, and changes from baseline at two years.
Mean Inspiratory and Expiratory Pressure (MIP/MEP) | Baseline and 2 years
  Static respiratory pressures at baseline, and changes from baseline at two years
Forced Vital Capacity (FVC) | Baseline and 2 years
  Dynamic spirometry while sitting, and supine when normal sitting. Baseline and changes from baseline at 2 years
Diaphragm thickness ratio | Baseline and 2 years
  Using ultrasound to measure thickness of diaphragm at maximum inspiration and at end-expiration. Ratio < 1,2 indicates reduced diaphragm movement. Bott left and right side will be measured.
Nocturnal oxygen saturation | Baseline and 2 years
  Monitor transcutaneous oxygen saturation during sleep.
Cough Peak Flow | Baseline and 2 years
  Cough Peak Flow at baseline and changes from baseline at 2 years
Apnea-hypopnea index | Baseline
  Using polysomnography to calculate the number of obstructive and non-obstructive apnea and hypopnea events pr hour sleep.
Respiratory disturbance index | Baseline
  Using polysomnography to calculate the number of respiratory events in terms of apneas, hypopneas and respiratory effort-related arousals pr hour sleep.
Thoracoabdominal breathing pattern during sleep | Baseline
  Using polysomnography to detect paradoxal breathing movements during sleep (abdomen moving in on inspiration when supine).
Echocardiography - conventional | Baseline and 2 years
  Measure cardiac function at baseline and changes from baseline at 2 years
Electrocardiography (ECG) | Baseline and 2 years
  Assessment of cardiac electrical activity at baseline and changes from baseline at 2 years
Pain (visual analogous scale, VAS) | Baseline and 2 years
  Patient-reported pain on VAS at baseline and at 2 years
Fatigue (Visual Analogous Scale, VAS) | Baseline and 2 years
  Patient-reported fatigue on VAS tat baseline and at 2 years
Fatigue Severity Scale (FSS) | Baseline and 2 years
  Fatigue at baseline and at 2 years
Epworth Sleepiness Scale (ESS) | Baseline
  Assessment of daytime sleepiness at baseline
Capillary blood gas | Baseline and 2 years
  Capillary CO2 at baseline and at 2 years
Serum Creatine Kinase (s-CK) | Baseline
  s-CK at baseline and at 2 years
Insomnia | Baseline
  Using Bergen Insomnia Scale to measure insomnia.
Sleep quality | Baseline
  Using Pittsburgh Sleep Quality index to measure sleep quality
Cognitive status | Baseline
  Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Arne Arntzen, ph.d, Principal Investigator — University Hospital of North Norway
Locations (1):
- National Neuromuscular Centre, Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No